CLINICAL TRIAL: NCT02631174
Title: Evaluation Of The Pharmacokinetics Of Antithrombin III In Neonates And Infants Undergoing CPB And ECMO Support
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014-6716
Record Dates: First submitted 2015-11-13; First posted 2015-12-16 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Extracorporeal Membrane Oxygenation Complication; Cardiopulmonary Bypass
MeSH Terms: interventions — Antithrombin III

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- cohort 1 (No Intervention): Cohort 1 (Aim 1) - 6 participants Cohort 1 will be comprised of 6 neonates (≤28 days of age) admitted to the CICU or NICU who are neither undergoing ECMO nor CPB. Cohort 1 will receive a single dose of ATIII by short 15 minute infusion.
- cohort 2.1 (Active Comparator): • Cohort 2.1 - 6 neonates undergoing ECMO.
  * Three participants will receive a single dose 15 minute infusion of hpATIII that is dose adjusted to account for additional circuit volume followed by a single dose 15 minute infusion of ATIII that is not dose adjusted to account for circuit volume
  * Three participants will receive a single dose 15 minute infusion of hpATIII that is not dose adjusted to account for circuit volume followed by a single dose 15 minute infusion of hpATIII that is dose adjusted to account for additional circuit volume
  Interventions: Drug: Antithrombin III
- cohort 2.2 (Active Comparator): • Cohort 2.2 - 12 neonates who will undergo open-heart surgery with CPB
  * Six participants will receive a single dose 15 minute infusion of ATIII that is dose adjusted to account for additional circuit volume.
  * Six participants will receive a single dose 15 minute infusion of ATIII that is not dose adjusted to account for circuit volume
  Interventions: Drug: Antithrombin III
- cohort 2.3 (Active Comparator): • Cohort 2.3 - 12 infants who will undergo open-heart surgery with CPB
  * Six participants will receive a single dose 15 minute infusion of ATIII that is dose adjusted to account for additional circuit volume.
  * Six participants will receive a single dose 15 minute infusion of ATIII that is not dose adjusted to account for circuit volume
  Interventions: Drug: Antithrombin III
- cohort 3 (Active Comparator): Cohort 3 (Aim 3) - 6 participants Six participants (neonates or infants) who will undergo ECMO and receive ATIII as standard of care will be enrolled and have a baseline ATIII level measured within 6 hours of ATIII administration and repeated within 15 minutes of initiation of extracorporeal support. If post-support level is < 80% normal activity then an ATIII level will be repeated and participants will be assigned to one of two hpATIII dosing regimens in which one formula accounts for additional circuit volume and one formula does not account for additional circuit volume, as described in section 7.4. Upon completion and 120 hr follow up after the first dose, participants still having ATIII activity less than 80% will then receive a second dose
  Interventions: Drug: Antithrombin III

INTERVENTIONS:
Drug: Antithrombin III — We are comparing neonates and infants on ECMP or CPB receiving ATIII, the dose of which is calculated to account for circuit volume, and compared with those not accounting for circuit volume
  Arms: cohort 2.1; cohort 2.2; cohort 2.3; cohort 3

SUMMARY:
The potential role of ATIII in achieving and maintaining adequate anticoagulation in pediatric patients on the heart-lung machine has recently taken on increased importance as caregivers strive to mitigate the risk for clinically significant clotting problems. It is known that ATIII levels are decreased in normal neonates and infants less than 6 months of age relative to older children and adults and become even further decreased in critically ill neonates and infants, including those with congenital heart disease. The current utilization of ATIII in the context of support on a heart-lung machine is based on pharmacokinetic data derived from adult subjects with congenital ATIII deficiency. There is a gap in knowledge as to the appropriate frequency of ATIII repletion, best method of monitoring, and mode of administration in critically ill neonates and infants receiving support on a heart-lung machine.Our long-term goal is to determine if antithrombin (ATIII) can effectively change the coagulation system in patients undergoing heart-lung machine support. The objective of this proposal, which is our first step in pursuit of that goal, is to determine the pharmacokinetics of ATIII in neonates and infants. Our central hypothesis is that ATIII will have different pharmacokinetic properties in neonates and infants than adults and these properties will be affected by the use of heart-lung machine.

This research will result in critical data on the pharmacokinetics of ATIII in neonates and infants receiving heart-lung machine support. This contribution is significant because it is the first step in a continuum of research that is expected to lead to the development of a therapeutic strategy employing ATIII that will facilitate improved modulation of the coagulation cascade to prevent significant clotting and bleeding complications in pediatric patients requiring heart-lung machine support.

DETAILED DESCRIPTION:
This is a single-site, prospective, open-label, pharmacokinetic study of hpATIII in neonates and infants. Patients admitted to the Cardiac Intensive Care Unit (CICU) and the Neonatal Intensive Care Unit (NICU) at Cincinnati Children's Hospital Medical Center (CCHMC) will be enrolled. Participants will be enrolled into one of three cohorts depending on whether they are scheduled for ECMO, CPB, or neither, and based on age (neonate or infant).

Two doses of hpATIII will be used; one according to current labelling for hpATIII and one that accounts for the additional circuit volume from ECMO or CPB. Pharmacokinetic measurements will be obtained for all groups at baseline prior to administration of hpATIII and at multiple defined times up to 120 hrs following each administration of hpATIII.

Administration of hpATIII is standard of care at CCHMC for participants undergoing ECMO. The standard dose administered for clinical care is (120 - baseline AT activity level) x weight (kg) / 1.4. For participants not undergoing ECMO for clinical care, or for those undergoing ECMO but receiving an adjusted dose for additional circuit volume , the administration of hpATIII is considered research.

The duration of the study at CCHMC is expected to be 2.5 years. This includes 24 months for recruitment and data collection, and 6 months for data analysis and report writing.

Individual participants will be in the study for approximately 120 hours (5 days) following administration of hpATIII. If participants receive more than 1 dose, they will be in the study for approximately 120 hours following each dose of hpATIII received.

ELIGIBILITY:
Inclusion Criteria:

* 1. Neonates less than or equal to 28 days of age OR Infants between 29 days and 1 year of age;
* 2. ATIII activity less than 80% at time of screening;

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from the study:

  1. Known or suspected bleeding disorder;
  2. Neonates with gestational age <36 weeks;
  3. Neonates with evidence of intracranial hemorrhage on routine cranial ultrasound;
  4. Documented infection (sepsis);
  5. Patients who require post-cardiotomy ECMO;
  6. Patients who require E-CPR; and/or
  7. Neonates or infants deemed to be at increased risk as judged by the investigator or for whom administration of hpATIII is not in their best interest
  8. Additional Exclusion for Cohort 1 only: Transfusion of whole blood, fresh frozen plasma (FFP), platelets or cryoprecipitate prior to study;

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2015-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Aim 1:To determine the pharmacokinetics of a single dose of hpATIII in neonates not undergoing ECMO or CPB. | participants in cohort 1 will have sampling up to 36 hrs after receiving their single dose of ATIII
  Blood samples (0.5 mL) for analysis of plasma ATIII concentration will be drawn at specific time points, e.g. before and after the dose of ATIII is given ,together with coagulation labs such as prothrombin/ thrombin anti thrombin complex and CBC, PT/PTT/INR at baseline, 12 and 24 hrs only.If clinical labs exist, those will be used instead for that time point.
Aim 2:To determine the pharmacokinetics of a single dose of hpATIII in neonates and infants undergoing ECMO or CPB | participants will be followed for 120hrs after recieving their single dose of ATIII
  Blood samples (0.5 mL) for analysis of plasma ATIII concentration will be drawn at specific time points, e.g.before and after the dose of ATIII is given,together with coagulation labs such as prothrombin/ thrombin anti thrombin complex and CBC, PT/PTT/INR at baseline, 12 and 24 hrs only. If clinical labs exist, those will be used instead for that time point.
Aim 3:To determine the pharmacokinetics of hpATIII administered by continuous infusion in neonates and infants undergoing ECMO | participants will be followed for a period of 120hrs after recieving half the dose as a bolus and the rest as a continuous infusion
  Blood samples (0.5 mL) for analysis of plasma ATIII concentration will be drawn at specific time points, e.g.before and after the dose of ATIII is given,together with coagulation labs such as prothrombin/ thrombin anti thrombin complex and CBC, PT/PTT/INR at baseline, 12 and 24 hrs only. If clinical labs exist, those will be used instead for that timepoint.

CONTACTS AND LOCATIONS:
Overall Officials: David Cooper, MD, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Guzzetta NA, Bajaj T, Fazlollah T, Szlam F, Wilson E, Kaiser A, Tosone SR, Miller BE. A comparison of heparin management strategies in infants undergoing cardiopulmonary bypass. Anesth Analg. 2008 Feb;106(2):419-25, table of contents. doi: 10.1213/01.ane.0000297290.03501.db. PMID 18227295
- [Background] D'Argenio DZ. Optimal sampling times for pharmacokinetic experiments. J Pharmacokinet Biopharm. 1981 Dec;9(6):739-56. doi: 10.1007/BF01070904. PMID 7341758
- [Background] Esmon CT. The interactions between inflammation and coagulation. Br J Haematol. 2005 Nov;131(4):417-30. doi: 10.1111/j.1365-2141.2005.05753.x. PMID 16281932
- [Background] Avidan MS, Levy JH, van Aken H, Feneck RO, Latimer RD, Ott E, Martin E, Birnbaum DE, Bonfiglio LJ, Kajdasz DK, Despotis GJ. Recombinant human antithrombin III restores heparin responsiveness and decreases activation of coagulation in heparin-resistant patients during cardiopulmonary bypass. J Thorac Cardiovasc Surg. 2005 Jul;130(1):107-13. doi: 10.1016/j.jtcvs.2004.10.045. PMID 15999048